CLINICAL TRIAL: NCT04032470
Title: Boston Scientific Registry of Deep Brain Stimulations for Treatment of Essential Tremor (ET):ET Registry
Brief Title: Boston Scientific Registry of Deep Brain Stimulation for Treatment of Essential Tremor (ET)
Status: Recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: A4080
Record Dates: First submitted 2019-07-08; First posted 2019-07-25 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Essential Tremor
Keywords: Deep Brain Stimulation; Boston Scientific; Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Essential Tremor: Subjects with Essential Tremor being implanted with Boston Scientific Deep Brain Stimulation Systems
  Interventions: Device: Deep Brain Stimulation Systems (DBS)

INTERVENTIONS:
Device: Deep Brain Stimulation Systems (DBS) — Subjects receiving DBS implant for treatment of Essential Tremor

SUMMARY:
To compile characteristics of real-world outcomes for Boston Scientific Corporation's commercially approved Deep Brain Stimulation (DBS) Systems, when used according to the applicable Directions for Use, for the treatment of Essential Tremor.

DETAILED DESCRIPTION:
To compile characteristics of real-world outcomes using Deep Brain Stimulation (DBS) for the treatment of Essential Tremor to add to the evidence available for treatment of ET.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria established in the locally applicable Directions for Use (DFU) for Essential Tremor
* Is at least 18 years old

Exclusion Criteria:

* Meets any contraindication in locally applicable Directions for Use

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with Essential Tremor
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-10-23 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life during the study as compared with baseline using the Quality of Life in Essential Tremor Questionnaire (QUEST) | Up to 3 years
  Change in quality of life over the course of the study using QUEST

OTHER OUTCOMES:
Change in tremor scores during the study as compared with baseline as assessed by Fahn-Tolosa- Marin Rating Scale | Up to 3 years
  Improvement in tremor scores as assessed by Fahn-Tolosa-Marin Tremor Rating Scale (FTMTRS) during the study as compared with baseline
Impression of Change scores during the study using Global Impression of Change | Up to 3 years
  Impression of Change scores during the study using Global Impression of Change

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bloom Lyons, Study Director — Boston Scientific Corporation
Locations (20):
- A.o. LKH Univ.-Kliniken Innsbruck, Innsbruck, Austria
- Belgium (3):
  - AZ Sint-Lucas, Ghent
  - UZ Gasthuisberg, Leuven
  - AZ Delta, Roeselare
- Vancouver General Hospital, Vancouver, Canada
- Germany (7):
  - Uniklinik Koln, Cologne
  - Universitaetsklinikum Dusseldorf, Düsseldorf
  - Universitaetsklinikum Essen, Essen
  - Universitatsklinikum Campus Kiel, Kiel
  - Universitaetsklinikum Giessen und Marburg GmbH, Marburg
  - Evangelisches Krankenhaus Oldenburg, Oldenburg
  - Universitaetsklinikum Wuerzburg, Würzburg
- Medical School of University PECS, Pécs, Hungary
- Policlinico Universitario Agostino Gemelli, Rome, Italy
- CHU Sao Joao, Porto, Portugal
- South Korea (3):
  - Samsung Medical Center, Seoul
  - Seoul ASAN Medical Center, Seoul
  - Yonsei University Severance Hospital, Seoul
- Spain (2):
  - Hospital De Bellvitge, Barcelona
  - Hospital General De Asturias, Oviedo